

# BROWN UNIVERSITY CONSENT FOR RESEARCH PARTICIPATION

Targeting Worry to Improve Sleep Version 3 – 7/5/19

## **KEY INFORMATION:**

You are invited to take part in a Brown University research study, which is being conducted at Brown in collaboration with Georgetown University. Your participation is voluntary.

- PURPOSE: The study is about seeing if an app-based mindfulness training program can help you decrease your worry and improve your sleep.
- PROCEDURES: You will be asked to complete four assessments; three will be in-person at Brown University and one will be completed online. You will also be asked to download and use the Unwinding Anxiety app on your phone on a daily basis. In addition, you will be asked to track your sleep for three, one week periods with a Fitbit Inspire & sleep diaries. You will also receive check-in phone calls.
- TIME INVOLVED: The first assessment will take  $\sim$ 1 hour to complete and the subsequent assessments will take  $\sim$ 45 minutes. In total the assessments will take approximately 3 hours and 30 minutes of your time. The daily app use will take approximately 10-15 minutes each day and you will be asked to complete the daily lesson once per day for 30 days.
- COMPENSATION: You will receive a \$25 Amazon gift card per assessment for a possible total of \$100 in Amazon gift cards. You will also receive lifetime access to the Unwinding Anxiety app and if you complete the entire study, you will get to keep the Fitbit Inspire.
- RISKS: 1) Loss of privacy protection: It is possible the data we collect could be lost or revealed. We will do everything we can to protect your privacy. 2) Possible side effects of using Unwinding Anxiety program: While we have not had reported side effects from this program, there have been some reports of side effects from other mindfulness meditation training interventions which will be described in more detail below. 3) Emotional distress from completing questionnaires: It is possible that you may experience temporary emotional distress as some of the questions are sensitive in nature.
- BENEFITS: There are no direct benefits to you for participating in this research study.
- ALTERNATIVES TO PARTICIPATION: Standard treatments for anxiety disorders include medication and talk therapy. Please contact your doctor for more information about anxiety treatments.

## 1. Researcher(s):

Principal Investigators: Judson Brewer, MD PhD, 401-863-2826 or judson\_brewer@brown.edu and Elizabeth Hoge, MD, 202-687-0635 or eah103@georgetown.edu

Project Coordinator: Alana Deluty, 401-297-0097, or Alana deluty@brown.edu (contact person).



## 2. What is this study about?

The purpose of this study is to see if an app, Unwinding Anxiety, (UA) can help decrease worry and improve sleep.

You are being asked to be in this study because you are over the age of 18, have a smartphone, and worry interferes with your ability to sleep.

#### 3. What will I be asked to do?

The study will consist of four assessments which are explained in more detail below.

Baseline, third, and fourth assessments (in-person)

## Questionnaires

During your first visit, you will be asked to complete several questionnaires which will cover a range of topics from demographic information, worry, body awareness, and sleep quality. This will take approximately 30 minutes.

## **Shape-matching task**

You will be presented with two shapes and you have to decide if they are the same shape. Sometimes a third "distractor" shape will be presented which you should ignore. This will take approximately 25 minutes.

Second assessment (online)

#### **Ouestionnaires**

You will complete several questionnaires pertaining to worry, body awareness, and sleep quality. This will take approximately 20 minutes.

In addition, you will be asked to keep a sleep diary of what time you go to bed and wake up and wear a sleep tracker for a one-week period after the baseline and before the third and fourth assessment.

This study has two different groups of research participants. To decide which group you will be in, we will use a method of chance. This method is like flipping a coin or rolling dice. The groups are explained in more detail below:

If you are randomized into Group A – You will be asked to complete the baseline, second (online), and third (in-person) assessments and then you will be asked to download the app. You will complete the introductory module ( $\sim$ 10-15 minutes) and an initial survey ( $\sim$ 10 minutes). You will then complete the 30-day Core Training program of Unwinding Anxiety ( $\sim$ 10–15 minutes/day). Sixty days after receiving the app you will be asked to return for a final in-person assessment.



You will be contacted for check-in calls regarding your experience with the app which will occur on day 7, 14, and 45. App usage will be monitored and you may receive an additional phone call to troubleshoot any problems.

If you are randomized into Group B – You will be asked to complete the baseline assessment and upon completion, you will be asked to download the app. You will complete the introductory module ( $\sim$ 10-15 minutes) and an initial survey ( $\sim$ 10 minutes). You will then complete the 30-day Core Training program of Unwinding Anxiety ( $\sim$ 10–15 minutes/day). You will be asked to complete the second assessment (online) when you reach module 14 (or one month after receiving the app) and the third assessment (inperson) when you reach module 30 (or 2 months after receiving the app). 120 days after receiving the app you will be asked to return for a final in-person assessment.

You will be contacted for check-ins regarding your experience with the app which will occur on day 7, 14, and 45. App usage will be monitored and you may receive an additional phone call to troubleshoot any problems.

Your participation in this study may last up to 120 days.

## 4. Will I be paid?

You will receive a \$25 Amazon gift card for each assessment you complete. If you complete all four assessments, you have the potential to receive a total of \$100 in Amazon gift cards. You will also receive lifetime access to the Unwinding Anxiety application and if you complete the entire study, you will get to keep the Fitbit Inspire. If you lose or damage the Fitbit Inspire, or if it is stolen, prior to completion of the study, you will not receive a new one and your participation in this study will end.

## 5. What are the risks?

There is a small risk that your personal information could be lost or exposed. This is very unlikely to happen and we will do everything in our power to make sure that your information is protected. Please note that any information you share on the online community is available to the public so use at your own discretion. Details below (part 7).

While we have not had report of side effects from this program "Unwinding Anxiety," there have been some reports of side effects from other mindfulness meditation training interventions. These rare side effects include trouble thinking clearly or making decisions, increased anxiety symptoms, repeated thoughts of a stressful experience from the past, irritability, trouble enjoying things that were previously enjoyable, feeling distant or cut off from people, difficulty sleeping, headaches and/or body pain, hearing sensitivity, feeling disconnected from everything, feeling negative emotions more strongly, feelings of distress. We will ask you about side effects from the program after completion

There is a small possibility that the questionnaires completed during the assessments may cause temporary emotional distress. You can skip any questions you do not feel comfortable answering and can stop study activities at any time.



#### 6. What are the benefits?

You may not directly benefit from being in this research study.

## 7. How will my information be protected?

All questionnaires will be recorded in a secure research database application and only the PI and members of research team will have access to it. Every participant will be given a number called a Participant ID and all data will be matched to the ID rather than identifiers. The study key matching the ID to identifiers will be saved in a secure, password-protected server (Stronghold) and only the PI and research team will have access to it. It will be kept for at least three years after the end of the study and then it will be destroyed. The research team will track the number of modules you complete through a password-protected server.

Signed and dated consent forms will be kept in a locked filing cabinet in a locked office on Brown University's campus which only study personnel will have access to. They will be maintained for at least three years after study completion.

The Unwinding Anxiety and Fitbit applications do collect data that will not be accessed by the researchers or used for research purposes. Please see the attached addenda (Fitbit Privacy Policy & Unwinding Anxiety Privacy Policy) for more details.

Brown University IRB and Georgetown University IRB staff and the National Institute of Health sometimes review studies like this one to make sure they are being done safely and correctly. If a review of this study takes place, your records may be examined. The reviewers will protect your confidentiality.

Anonymized data may be used and/or shared for future research.

Certificate of Confidentiality: To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

The Certificate of Confidentiality will not be used to prevent disclosure to state or local authorities of child abuse and neglect, or harm to self or others.



Clinical Trial: A description of this clinical trial will be available on http://www.Clinical Trials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### 8. Are there any alternatives to this study?

Standard therapy for anxiety includes medications (such as selection serotonin-reuptake inhibitors) and behavioral treatments (such as cognitive behavioral therapy). You can contact your doctor for more information. In addition, a resource/referral list will be provided after reviewing the consent form.

## 9. What if I want to stop?

You do not have to be in this study if you do not want to be. Even if you decide to be in this study, you can change your mind and stop at any time.

If you refuse to participate in or leave the study, your current or future relationships with Brown University and Georgetown University will not be affected. You will be asked to return the Fitbit Inspire at a time convenient to you.

## 10. What are the financial interests in this study?

You are being given this information so that you can decide if this relationship affects whether you want to participate in this study. If you have any questions, please contact Project Coordinator: Alana Deluty, 401-297-0097, or Alana deluty@brown.edu (contact person). They will answer any questions you may have.

Dr. Brewer is the lead researcher in this study and is one of the founders of, and has equity in, MindSciences, the company that created the Unwinding Anxiety app being studied. He may benefit financially if the Unwinding Anxiety program is successful.

Dr. Brewer will not be enrolling or consenting participants. Any publication of this study will require a statistician independent of the study and Mindsciences. Dr. Brewer will disclose his relationship to the company in any publications or presentations about this study.

## 11. Who can I talk to if I have questions about this study?

If you have any questions about your participation in this study, you can call Project Coordinator: Alana Deluty, 401-297-0097, or Alana\_deluty@brown.edu (contact person). You can also call the Principal Investigator, Judson Brewer, MD PhD at 401-863-2826 or email him at Judson\_brewer@brown.edu.

## 12. Who can I talk to if I have questions about my rights as a participant?



If you have questions about your rights as a research participant, you can contact Brown University's Human Research Protection Program at 401-863-3050 or email them at <a href="mailto:IRB@Brown.edu">IRB@Brown.edu</a>.

## 13. Future Studies

| There are other studies that I may be eligible for in the future. The Mindfulness Center at Brown University may contact me to invite me to participate in other research studies if I check the box below. I would like the Mindfulness Center at Brown University to invite me to participate in other research studies. | | |
|---|---|---|
| Your signature below shows that you he that you agree to volunteer as a research | | understood the information in this document, and for this study. |
| You will be offered a copy of this form | | |
| Participant's Signature and Date | / | PRINTED NAME |
| Research Staff Signature and Date | / | PRINTED NAME |

## Addendum A – Fitbit Privacy Policy

## Specifically, we'll cover:

- Information We Collect
- How We Use Information
- How Information Is Shared
- Your Rights To Access and Control Your Personal Data
- Data Retention
- Information Security
- Who We Are and How To Contact Us

## INFORMATION WE COLLECT

When you use our Services, we collect the following types of information.

## INFORMATION YOU PROVIDE US

## ACCOUNT INFORMATION

Some information is required to create an account on our Services, such as your name, email address, password, date of birth, gender, height, weight, and in some cases your mobile telephone number. This is the only information you have to provide to create an account with us. You may also choose to provide other types of information, such as a profile photo, biography, country information, and community username.

#### ADDITIONAL INFORMATION

To help improve your experience or enable certain features of the Services, you may choose to provide us with additional information, like your logs for food, weight, sleep, water, or female health tracking; an alarm; and messages on discussion boards or to your friends on the Services.

You may also connect with friends on the Services or invite friends who have not yet joined by providing their email addresses, accessing social networking accounts, or using the contact list on your mobile device. We do not store your contact list and delete it after it is used for adding contacts as friends.

If you contact us or participate in a survey, contest, or promotion, we collect the information you submit such as your name, contact information, and message.

## PAYMENT AND CARD INFORMATION

Some Fitbit devices support payments and transactions with third parties. If you activate this feature, you must provide certain information for identification and verification, such as your name, credit, debit or other card number, card expiration date, and CVV code. This information is encrypted and sent to your card network, which upon approval sends back to your device a token, which is a set of random digits for engaging in transactions without exposing your card number. For your convenience, we store the last four digits of your card number and your card issuer's name and contact information. You can remove the token from your account using your account settings. We do not store your transaction history.

If you purchase Fitbit merchandise on our website, you provide your payment information, including your name, credit or debit card number, card expiration date, CVV code, and billing address. We do not store this payment information. We store your shipping address to fulfill your order. Note that third-party payment processors may retain this information in accordance with their own privacy policies and terms.

#### LIVE COACHING SERVICES

Our live coaching services are a platform for you to communicate with a live health, fitness, or wellness coach ("Live Coaching Services"). Coaches may be provided by third parties, such as your employer or insurance company, or by our third-party coaching service providers. If you use our Live Coaching Services, we collect information about such use, including the plan, goals, and actions you record with your coach, your calendar events, communications with your coach, notes your coach records about you, and other information submitted by you or your coach.

## INFORMATION WE RECEIVE FROM YOUR USE OF OUR SERVICES

#### **DEVICE INFORMATION**

Your device collects data to estimate a variety of metrics like the number of steps you take, your distance traveled, calories burned, weight, heart rate, sleep stages, active minutes, and location. The data collected varies depending on which device you use. Learn more about the features of <u>our various devices</u> and how you can use <u>MobileTrack</u>. When your device syncs with our applications or software, data recorded on your device is transferred from your device to our servers.

## LOCATION INFORMATION

The Services include features that use precise location data, including GPS signals, device sensors, Wi-Fi access points, and cell tower IDs. We collect this type of data if you grant us access to your location. You can always remove our access using your Fitbit device or mobile device settings. We may also derive your approximate location from your IP address.

#### USAGE INFORMATION

When you access or use our Services, we receive certain usage data. This includes information about your interaction with the Services, for example, when you view or search content, install applications or software, create or log into your account, pair your device to your account, or open or interact with an application on your Fitbit device.

We also collect data about the devices and computers you use to access the Services, including IP addresses, browser type, language, operating system, Fitbit or mobile device information (including device and application identifiers), the referring web page, pages visited, location (depending on the permissions you have granted us), and cookie information.

## INFORMATION WE RECEIVE FROM THIRD PARTIES

If you choose to connect your account on our Services to your account on another service, we may receive information from the other service. For example, if you connect to Facebook or Google, we may receive information like your name, profile picture, age range, language, email address, and friend list. You may also choose to grant us access to your exercise or activity data from another service. You can stop sharing the information from the other service with us by removing our access to that other service.

We may partner with third parties, such as employers and insurance companies that offer Fitbit services to their employees and customers. In such cases, those companies may provide us with your name, email address, or similar information (like a telephone number or subscriber ID) so that we can invite you to participate or determine your eligibility for particular benefits, such as discounts or free services.

## HEALTH AND OTHER SPECIAL CATEGORIES OF PERSONAL DATA

To the extent that information we collect is health data or another special category of personal data subject to the European Union's General Data Protection Regulation ("GDPR"), we ask for your explicit consent to process the data. We obtain this consent separately when you take actions leading to our obtaining the data, for example, when you pair your device to your account, grant us access to your exercise or activity data from another service, or use the female health tracking feature. You can use your account settings and tools to withdraw your consent at any time, including by stopping use of a feature, removing our access to a third-party service, unpairing your device, or deleting your data or your account.

## HOW WE USE INFORMATION

We use the information we collect for the following purposes.

#### PROVIDE AND MAINTAIN THE SERVICES

Using the information we collect, we are able to deliver the Services to you and honor our <u>Terms of Service</u> contract with you. For example, we need to use your information to provide you with your Fitbit dashboard tracking your exercise, activity, and other trends; to enable the community features of the Services; and to give you customer support.

For the Services' community features, we may use your information to help you find and connect with other users and to allow other users to find and connect with you. For example, your account contact information allows other users to add you as a friend. When another user has your email or mobile phone number in their contact list or in their friend network on a connected service, we show that user that you are a user of the Services.

If you use the Live Coaching Services, we use your information to connect you with coaches, allow you to communicate with them through our Services, and help you achieve your goals to lead a healthier, more active life. For example, the goals that you provide allow you to develop a personal plan and set of actions in consultation with your coach.

## IMPROVE, PERSONALIZE, AND DEVELOP THE SERVICES

We use the information we collect to improve and personalize the Services and to develop new ones. For example, we use the information to troubleshoot and protect against errors; perform data analysis and testing; conduct research and surveys; and develop new features and Services.

When you allow us to collect precise location information, we use that information to provide and improve features of the Services such as recording where a workout took place or mapping an activity.

We also use your information to make inferences and show you more relevant content. Here are some examples:

- Information like your height, weight, gender, and age allows us to improve the accuracy of your daily exercise and activity statistics like the number of calories you burned and the distance you traveled.
- Based on your sleep data, we may make inferences about your sleeping patterns and provide you with customized insights to help you improve your sleep.
- We may personalize exercise and activity goals for you based on the goals you previously set and your historical exercise or activity data.

## **COMMUNICATE WITH YOU**

We use your information when needed to send you Service notifications and respond to you when you contact us. We also use your information to promote new features or products that we think you would be interested in. You can control marketing communications and most Service notifications by using your <u>notification</u> <u>preferences</u> in <u>account settings</u> or via the "Unsubscribe" link in an email.

## PROMOTE SAFETY AND SECURITY

We use the information we collect to promote the safety and security of the Services, our users, and other parties. For example, we may use the information to authenticate users, facilitate secure payments, protect against fraud and abuse, respond to a legal request or claim, conduct audits, and enforce our terms and policies.

We use cookies and similar technologies for the purposes described above. For more information, please read our Cookie Use statement.

For personal data subject to the GDPR, we rely on several legal bases to process the data. These include when you have given your consent, which you may withdraw at any time using your <u>account settings</u> and other tools; when the processing is necessary to perform a contract with you, like the <u>Terms of Service</u>; and our legitimate business interests, such as in improving, personalizing, and developing the Services, marketing new features or products that may be of interest, and promoting safety and security as described above.

## HOW INFORMATION IS SHARED

We do not share your personal information except in the limited circumstances described below.

#### WHEN YOU AGREE OR DIRECT US TO SHARE

You may direct us to disclose your information to others, such as when you use our community features like the forums, 7-day leaderboard, and other social tools. For certain information, we provide you with <u>privacy preferences</u> in <u>account settings</u> and other tools to control how your information is visible to other users of the Services. Just remember that if you choose to participate in a challenge, information like your profile photo, posted messages, total steps in the challenge, personal statistics, and achievements, is not governed by your <u>privacy preferences</u> and will be visible to all other challenge participants.

You may also authorize us to share your information with others, for example, with a third-party application when you give it access to your account, or with your employer when you choose to participate in an employee wellness program. Remember that their use of your information will be governed by their privacy policies and terms. You can revoke your consent to share with third-party applications or employee wellness programs using your account settings.

## FOR EXTERNAL PROCESSING

We transfer information to our corporate affiliates, service providers, and other partners who process it for us, based on our instructions, and in compliance with this policy and any other appropriate confidentiality and security measures. These partners provide us with services globally, including for customer support, information technology, payments, sales, marketing, data analysis, research, and surveys.

#### FOR LEGAL REASONS OR TO PREVENT HARM

We may preserve or disclose information about you to comply with a law, regulation, legal process, or governmental request; to assert legal rights or defend against legal claims; or to prevent, detect, or investigate illegal activity, fraud, abuse, violations of our terms, or threats to the security of the Services or the physical safety of any person.

Please note: Our policy is to notify you of legal process seeking access to your information, such as search warrants, court orders, or subpoenas, unless we are prohibited by law from doing so. In cases where a court order specifies a non-disclosure period, we provide delayed notice after the expiration of the non-disclosure period. Exceptions to our notice policy include exigent or counterproductive circumstances, for example, when there is an emergency involving a danger of death or serious physical injury to a person.

We may share non-personal information that is aggregated or de-identified so that it cannot reasonably be used to identify an individual. We may disclose such information publicly and to third parties, for example, in public reports about exercise and activity, to partners under agreement with us, or as part of the community benchmarking information we provide to users of our subscription services.

If we are involved in a merger, acquisition, or sale of assets, we will continue to take measures to protect the confidentiality of personal information and give affected users notice before transferring any personal information to a new entity.

## YOUR RIGHTS TO ACCESS AND CONTROL YOUR PERSONAL DATA

We give you <u>account settings</u> and tools to access and control your personal data, as described below, regardless of where you live. If you live in the European Economic Area, United Kingdom, and Switzerland (the "Designated Countries"), you have a number of legal rights with respect to your information, which your <u>account settings</u> and tools allow you to exercise, as outlined below.

Accessing and Exporting Data. By logging into your account, you can access much of your personal information, including your dashboard with your daily exercise and activity statistics. Using your <u>account settings</u>, you can also download information in a commonly used file format, including data about your activities, body, foods, and sleep.

Editing and Deleting Data. Your <u>account settings</u> let you change and delete your personal information. For instance, you can edit or delete the profile data you provide and delete your account if you wish. If you choose to delete your account, please note that while most of your information will be deleted within 30 days, it may take up to 90 days to delete all of your information, like the data recorded by your Fitbit device and other data stored in our backup systems. This is due to the size and complexity of the systems we use to store data. We may also preserve data for legal reasons or to prevent harm, including as described in the <u>How Information Is Shared</u> section.

Objecting to Data Use. We give you <u>account settings</u> and tools to control our data use. For example, through your <u>privacy settings</u>, you can limit how your information is visible to other users of the Services; using your <u>notification settings</u>, you can limit the notifications you receive from us; and under your <u>application settings</u>, you can revoke the access of third-party applications that you previously connected to your Fitbit account. You can also use the Fitbit application to unpair your device from your account at any time.

If you live in a Designated Country, in certain circumstances, you can object to our processing of your information based on our legitimate interests, including as described in the <a href="How We Use Information">How We Use Information</a> section. You have a general right to object to the use of your information for direct marketing purposes. Please see your <a href="notification settings">notification settings</a> to control our marketing communications to you about Fitbit products. Please also review our <a href="Cookie Use">Cookie Use</a> statement for your options to control how we and our partners use cookies and similar technologies for advertising.

Restricting or Limiting Data Use. In addition to the various controls that we offer, if you reside in a Designated Country, you can seek to restrict our processing of your data in certain circumstances. Please note that you can always delete your account at any time.

If you need further assistance regarding your rights, please contact our Data Protection Officer at <a href="mailto:data-protection-office@fitbit.com">data-protection-office@fitbit.com</a>, and we will consider your request in accordance with applicable laws. If you reside in a Designated Country, you also have a right to lodge a complaint with your local data protection authority or with the Irish Data Protection Commissioner, our lead supervisory authority, whose contact information is available here.

## DATA RETENTION

We keep your account information, like your name, email address, and password, for as long as your account is in existence because we need it to operate your account. In some cases, when you give us information for a feature of the Services, we delete the data after it is no longer needed for the feature. For instance, when you provide your contact list for finding friends on the Services, we delete the list after it is used for adding contacts as friends. We keep other information, like your exercise or activity data, until you use your account settings or tools to delete the data or your account because we use this data to provide you with your personal statistics and other aspects of the Services. We also keep information about you and your use of the Services for as long as necessary for our legitimate business interests, for legal reasons, and to prevent harm, including as described in the <a href="How We Use Information">How Information Is Shared</a> sections.

## INFORMATION SECURITY

We work hard to keep your data safe. We use a combination of technical, administrative, and physical controls to maintain the security of your data. This includes using Transport Layer Security ("TLS") to encrypt many of our Services. No method of transmitting or storing data is completely secure, however. If you have a security-related concern, please contact <u>Customer Support</u>.

## <u>Addendum B – Mindsciences Privacy Policy</u>

Effective date: September 26, 2018

MindSciences, Inc. ("us", "we", or "our") operates

the https://www.drjud.com,https://www.mindsciences.com, http://www.unwindinganxie ty.com, http://www.goeatrightnow.com, and http://www.cravingtoquit.com websites and the Unwinding Anxiety, Eat Right Now, and Craving to Quit programs, including related mobile applications and online Communities (hereinafter referred to as the "Services"). This page informs you of our policies regarding the collection, use and disclosure of personal data when you use our Services and the choices you have associated with that data.

We use your data to provide and improve the Services. By using the Services, you agree to the collection and use of information in accordance with this policy. Unless otherwise defined in this Privacy Policy, the terms used in this Privacy Policy have the same meanings as in our Terms and Conditions.

#### **Definitions**

#### **Services**

Services means

the https://www.drjud.com, https://www.mindsciences.com,http://www.unwindinganxie ty.com, http://www.goeatrightnow.com, andhttp://www.cravingtoquit.com websites and the Unwinding Anxiety, Eat Right Now, and Craving to Quit programs, including related mobile applications and online Communities operated by MindSciences, Inc.

#### Personal Data

Personal Data means data about a living individual who can be identified from those data

#### **Usage Data**

Usage Data is data collected automatically either generated by the use of the Services or from the Services infrastructure itself (for example, the duration of a page visit).

## **Cookies**

Cookies are small files stored on your device (computer or mobile device).

## **Data Controller**

Data Controller means the natural or legal person who (either alone or jointly or in common with other persons) determines the purposes for which and the manner in which any personal information are, or are to be, processed.

For the purpose of this Privacy Policy, we are a Data Controller of your Personal Data.

## **Data Processors (or Services Providers)**

Data Processor (or Services Provider) means any natural or legal person who processes the data on behalf of the Data Controller.

We may use the Services of various Services Providers in order to process your data more effectively.

## Data Subject (or User)

Data Subject is any living individual who is using our Services and is the subject of Personal Data.

#### **Information Collection and Use**

We collect several different types of information for various purposes to provide and improve our Services to you. If you subscribe to the Products as part of a 3rd party program, for example, but not limited to, an insurer or benefits supplier, MindSciences may share all data it has with that 3rd party.

## **Types of Data Collected**

#### **Personal Data**

While using our Services, we may ask you to provide us with certain personally identifiable information that can be used to contact or identify you ("Personal Data"). Personally identifiable information may include:

- Email address
- First name and last name
- Phone number
- Address, State, Province, ZIP/Postal code, City
- Cookies and Usage Data

We may use your Personal Data to contact you with newsletters, marketing or promotional materials and other information that may be of interest to you. You may opt out of receiving any, or all, of these communications from us by following the unsubscribe link or the instructions provided in any email we send.

## **Usage Data**

We may also collect information that your browser sends whenever you visit our Services or when you access the Services by or through a mobile device ("Usage Data").

This Usage Data may include information such as your computer's Internet Protocol address (e.g. IP address), browser type, browser version, the pages of our Services that you

visit, the time and date of your visit, the time spent on those pages, unique device identifiers and other diagnostic data.

When you access the Services with a mobile device, this Usage Data may include information such as the type of mobile device you use, your mobile device unique ID, the IP address of your mobile device, your mobile operating system, the type of mobile Internet browser you use, unique device identifiers and other diagnostic data.

#### **Tracking Cookies Data**

We use cookies and similar tracking technologies to track the activity on our Services and we hold certain information.

Cookies are files with a small amount of data which may include an anonymous unique identifier. Cookies are sent to your browser from a website and stored on your device. Other tracking technologies are also used such as beacons, tags and scripts to collect and track information and to improve and analyze our Services.

You can instruct your browser to refuse all cookies or to indicate when a cookie is being sent. However, if you do not accept cookies, you may not be able to use some portions of our Services.

Examples of Cookies we use:

- **Session Cookies.** We use Session Cookies to operate our Services.
- **Preference Cookies.** We use Preference Cookies to remember your preferences and various settings.
- **Security Cookies.** We use Security Cookies for security purposes.

#### **Use of Data**

MindSciences, Inc. uses the collected data for various purposes:

- To provide and maintain our Services
- To notify you about changes to our Services
- To allow you to participate in interactive features of our Services when you choose to do so
- To provide customer support
- To gather analysis or valuable information so that we can improve our Services
- To delelop new Products
- To conduct research and publish results
- To monitor the usage of our Services
- To detect, prevent and address technical issues
- To provide you with news, special offers and general information about other goods, Services and events which we offer that are similar to those that you have already purchased or enquired about unless you have opted not to receive such information

# Legal Basis for Processing Personal Data under the General Data Protection Regulation (GDPR)

If you are from the European Economic Area (EEA), MindSciences, Inc. legal basis for collecting and using the personal information described in this Privacy Policy depends on the Personal Data we collect and the specific context in which we collect it.

MindSciences, Inc. may process your Personal Data because:

- We need to perform a contract with you
- You have given us permission to do so
- The processing is in our legitimate interests and it is not overridden by your rights
- For payment processing purposes
- To comply with the law

#### **Retention of Data**

MindSciences, Inc. will retain your Personal Data only for as long as is necessary for the purposes set out in this Privacy Policy. We will retain and use your Personal Data to the extent necessary to comply with our legal obligations (for example, if we are required to retain your data to comply with applicable laws), resolve disputes and enforce our legal agreements and policies. Name and Email address will be retained for the purposes of contacting you regarding Products

MindSciences, Inc. will also retain Usage Data for internal analysis purposes.

#### **Transfer of Data**

Your information, including Personal Data, may be transferred to — and maintained on — computers located outside of your state, province, country or other governmental jurisdiction where the data protection laws may differ from those of your jurisdiction.

If you are located outside United States and choose to provide information to us, please note that we transfer the data, including Personal Data, to United States and process it there.

Your consent to this Privacy Policy followed by your submission of such information represents your agreement to that transfer.

MindSciences, Inc. will take all the steps reasonably necessary to ensure that your data is treated securely and in accordance with this Privacy Policy and no transfer of your Personal Data will take place to an organisation or a country unless there are reasonable controls in place including the security of your data and other personal information.

#### **Disclosure of Data**

#### **Business Transaction**

If MindSciences, Inc. is involved in a merger, acquisition or asset sale, your Personal Data may be transferred. We will provide notice before your Personal Data is transferred and becomes subject to a different Privacy Policy.

#### **Disclosure for Law Enforcement**

Under certain circumstances, MindSciences, Inc. may be required to disclose your Personal Data if required to do so by law or in response to valid requests by public authorities (e.g. a court or a government agency).

## **Legal Requirements**

MindSciences, Inc. may disclose your Personal Data in the good faith belief that such action is necessary to:

- To comply with a legal obligation
- To protect and defend the rights or property of MindSciences, Inc.
- To prevent or investigate possible wrongdoing in connection with the Services
- To protect the personal safety of users of the Services or the public
- To protect against legal liability

#### **Security of Data**

The security of your data is important to us but remember that no method of transmission over the Internet or method of electronic storage is 100% secure. While we strive to use commercially acceptable means to protect your Personal Data, we cannot guarantee its absolute security.

# Our Policy on "Do Not Track" Signals under the California Online Protection Act (CalOPPA)

We do not support Do Not Track ("DNT"). Do Not Track is a preference you can set in your web browser to inform websites that you do not want to be tracked.

You can enable or disable Do Not Track by visiting the Preferences or Settings page of your web browser.

## Your Data Protection Rights under the General Data Protection Regulation (GDPR)

If you are a resident of the European Economic Area (EEA), you have certain data protection rights. MindSciences, Inc. aims to take reasonable steps to allow you to correct, amend, delete or limit the use of your Personal Data.

If you wish to be informed about what Personal Data we hold about you and if you want it to be removed from our systems, please contact us.

In certain circumstances, you have the following data protection rights:

- The right to access, update or delete the information we have on you. Whenever made possible, you can access, update or request deletion of your Personal Data directly within your account settings section. If you are unable to perform these actions yourself, please contact us to assist you.
- The right of rectification. You have the right to have your information rectified if that information is inaccurate or incomplete.
- The right to object. You have the right to object to our processing of your Personal Data.
- The right of restriction. You have the right to request that we restrict the processing of your personal information.
- The right to data portability. You have the right to be provided with a copy of the information we have on you in a structured, machine-readable and commonly used format.
- The right to withdraw consent. You also have the right to withdraw your consent at any time where MindSciences, Inc. relied on your consent to process your personal information.

Please note that we may ask you to verify your identity before responding to such requests.

You have the right to complain to a Data Protection Authority about our collection and use of your Personal Data. For more information, please contact your local data protection authority in the European Economic Area (EEA).

#### **Services Providers**

We may employ third party companies and individuals to facilitate our Services ("Services Providers"), provide the Services on our behalf, perform Services-related Services or assist us in analysing how our Services is used.

These third parties have access to your Personal Data only to perform these tasks on our behalf and are obligated not to disclose or use it for any other purpose.

#### **Analytics**

We may use third-party Services Providers to monitor and analyze the use of our Services.

## Google Analytics

Google Analytics is a web analytics Services offered by Google that tracks and reports website traffic. Google uses the data collected to track and monitor the use of our Services. This data is shared with other Google Servicess. Google may use the collected data to contextualise and personalise the ads of its own advertising network.

For more information on the privacy practices of Google, please visit the Google Privacy Terms web page: https://policies.google.com/privacy?hl=en

#### Mixpanel

Mixpanel is provided by Mixpanel Inc.

You can prevent Mixpanel from using your information for analytics purposes by opting-out. To opt-out of Mixpanel Services, please visit this

page: https://mixpanel.com/optout/

For more information on what type of information Mixpanel collects, please visit the Terms of Use page of Mixpanel: https://mixpanel.com/terms/

## Other third-party Services Providers

From time to time we may use other third-party Services Providers to monitor and analyze the use of our Services.

## **Behavioral Remarketing**

MindSciences, Inc. uses remarketing Services to advertise on third party websites to you after you visited our Services. We and our third-party vendors use cookies to inform, optimise and serve ads based on your past visits to our Services.

## Google Ads (AdWords)

Google Ads (AdWords) remarketing Services is provided by Google Inc.

You can opt-out of Google Analytics for Display Advertising and customise the Google Display Network ads by visiting the Google Ads Settings page: http://www.google.com/settings/ads

Google also recommends installing the Google Analytics Opt-out Browser Add-on – https://tools.google.com/dlpage/gaoptout – for your web browser. Google Analytics Opt-out Browser Add-on provides visitors with the ability to prevent their data from being collected and used by Google Analytics.

For more information on the privacy practices of Google, please visit the Google Privacy Terms web page: https://policies.google.com/privacy?hl=en

## • Twitter

Twitter remarketing Services is provided by Twitter Inc.

You can opt-out from Twitter's interest-based ads by following their instructions:https://support.twitter.com/articles/20170405

You can learn more about the privacy practices and policies of Twitter by visiting their Privacy Policy page: https://twitter.com/privacy

#### Facebook

Facebook remarketing Services is provided by Facebook Inc.

You can learn more about interest-based advertising from Facebook by visiting this page:https://www.facebook.com/help/164968693837950

To opt-out from Facebook's interest-based ads, follow these instructions from Facebook:https://www.facebook.com/help/568137493302217

Facebook adheres to the Self-Regulatory Principles for Online Behavioural Advertising established by the Digital Advertising Alliance. You can also opt-out from Facebook and other participating companies through the Digital Advertising Alliance in the USAhttp://www.aboutads.info/choices/, the Digital Advertising

Alliance of Canada in Canadahttp://youradchoices.ca/ or the European Interactive Digital Advertising Alliance in Europehttp://www.youronlinechoices.eu/, or opt-out using your mobile device settings.

For more information on the privacy practices of Facebook, please visit Facebook's Data Policy:https://www.facebook.com/privacy/explanation

• Other third-party Services Providers:
From time to time we may use other third-party Services Providers to advertise.

## **Payments**

We may provide paid products and/or Services within the Services. In that case, we use third-party Services for payment processing (e.g. payment processors).

We will not store or collect your payment card details. That information is provided directly to our third-party payment processors whose use of your personal information is governed by their Privacy Policy. These payment processors adhere to the standards set by PCI-DSS as managed by the PCI Security Standards Council, which is a joint effort of brands like Visa, MasterCard, American Express and Discover. PCI-DSS requirements help ensure the secure handling of payment information.

The payment processors we work with are:

- Apple Store In-App Payments
   Their Privacy Policy can be viewed at https://www.apple.com/legal/privacy/en-ww/
- Google Play In-App Payments
  Their Privacy Policy can be viewed at https://www.google.com/policies/privacy/
- **Stripe**Their Privacy Policy can be viewed at https://stripe.com/us/privacy

#### **Links to Other Sites**

Our Services may contain links to other sites that are not operated by us. If you click a third-party link, you will be directed to that third party's site. We strongly advise you to review the Privacy Policy of every site you visit.

We have no control over and assume no responsibility for the content, privacy policies or practices of any third party sites or Services.

## **Children's Privacy**

Our Services does not address anyone under the age of 18 ("Children").

We do not knowingly collect personally identifiable information from anyone under the age of 18. If you are a parent or guardian and you are aware that your Child has provided us with Personal Data, please contact us. If we become aware that we have collected Personal

Data from children without verification of parental consent, we take steps to remove that information from our servers.

## **Changes to This Privacy Policy**

We may update our Privacy Policy from time to time. We will notify you of any changes by posting the new Privacy Policy on this page.

We will let you know via email and/or a prominent notice on our Services, prior to the change becoming effective and update the "effective date" at the top of this Privacy Policy.

You are advised to review this Privacy Policy periodically for any changes. Changes to this Privacy Policy are effective when they are posted on this page.

#### **Contact Us**

If you have any questions about this Privacy Policy, please contact us:

By email: support@mindsciences.com